CLINICAL TRIAL: NCT00513240
Title: Erythropoetin Neuroprotection for Neonatal Cardiac Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Dana Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dean Andropoulos, Professor, Chief of Pediatric Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R21HD5550101; IND #100011 (Other: FDA); 0942 (Other Grant/Funding Number: Baylor College of Medicine General Clinical Research Center); 1R21HD055501-01 (NIH); Not Assigned (Other Grant/Funding Number: Charles A. Dana Foundation Brain and Immuno-Imaging Grant)
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Congenital Heart Disease; Hypoplastic Left Heart Syndrome; Transposition of the Great Arteries; Aortic Arch Hypoplasia or Interruption
Keywords: erythropoetin; neuroprotection; neonate; cardiac; magnetic resonance imaging; brain magnetic resonance imaging; electroencephalogram
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Transposition of Great Vessels | interventions — Erythropoietin; Epoetin Alfa; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPO group (Experimental): Patients randomized to receive the 3 doses of erythropoetin.
  Interventions: Drug: Erythropoetin
- Control group. (Placebo Comparator): Patients randomized to receive 3 doses of normal saline control.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Erythropoetin — Erythropoetin 500 units/kg IV x 3 : dose 1. 12-72 hours preoperatively, dose 2. Postoperative day #1, 48 hours after separating from cardiopulmonary bypass, and dose 3. postoperative day #3, 48 hours after dose #2
  Other Names: Procrit; Epoetin alpha
  Arms: EPO group
Drug: Normal saline — Normal saline placebo in 3 doses:dose 1. 12-72 hours preoperatively, dose 2. Postoperative day #1, 48 hours after separating from cardiopulmonary bypass, and dose 3. postoperative day #3, 48 hours after dose #2.
  .
  Other Names: Saline placebo
  Arms: Control group.

SUMMARY:
Brain problems occur in neonatal open heart surgery with a frequency of 20-70%, seen on neurological examination, brain imaging such as magnetic resonance imaging (MRI), or long term development problems such as learning disorders and hyperactivity syndromes. This study aims to determine if erythropoetin, a natural hormone made in the body, protects the brain from damage when given in high doses before and during neonatal open heart surgery. We will use brain MRI, brain wave tests (EEG), neurological examination, and long term developmental outcome testing to see if erythropoetin is better than salt water injection (placebo) in protecting the brain.

DETAILED DESCRIPTION:
Hypothesis: Erythropoetin (EPO) will protect the neonatal brain in the perioperative period for congenital heart surgery.

Using a prospective, randomized, placebo-controlled, double-blinded design, the specific aims of this study are:

1. To determine the effect of perioperative EPO on short and long term neurological outcomes in neonates undergoing cardiac surgery with an optimized cardiopulmonary bypass strategy.
2. To determine EPO tolerability and safety with short term administration.
3. To determine EPO pharmacokinetics in this population.
4. To determine the relationship of neurological monitoring, specifically NIRS, to neurological outcomes with an optimized cardiopulmonary bypass technique in neonates that avoids deep hypothermic circulatory arrest, and to determine if EPO affects this relationship.

Protocol: Neonates undergoing arterial switch, Norwood, or aortic arch advancement/other complete 2 ventricle repair, >35 weeks gestation and ≥2.0 kg are eligible.

Preop day 1:NIRS for 12-24 hours, neuro exam, and Study drug dose #1: EPO 500 units/kg or saline placebo 12-72 hours before surgery. EPO Pharmacokinetic data for 25-50 consenting patients.

Day of surgery: Brain MRI immediately preop. Anesthesia/CPB per our standard practice (fentanyl 100-200 mcg/kg, midazolam, isoflurane, epsilon-aminocaproic acid, 75 mg/kg IV load to patient and CPB prime, and 75 mg/kg/hr infusion in OR) with ACP guided by TCD, pH stat, hct 30-35, avoid DHCA.

POD #1: Study drug dose #2: EPO 500 units/kg or saline placebo 24 hours after dose #2.

For 72 hours postop, NIRS monitoring. All monitor data collected electronically.

POD #3: Study drug dose #3: EPO 500 units/kg or saline placebo 48 hours after dose #3.

7 days postop: Brain MRI. (pentobarbital IV). Neuro exam before discharge. 3-6 months: Brain MRI immediately before or after 2nd surgery, or as outpatient (IV pentobarb or propofol/midazolam-may use N2O/sevo for induction, cannot intubate if outpatient; OR if cardiac MRI at same time, any indicated anesthetic technique). NIRS x 24h after 2nd surgery.

1,and 3 years: Bayley Scales of Infant Development III. 5 years: Battery of neurodevelopmental tests.

Early primary outcome variable: MRI severity of injury score (decrease by 25%). Late outcome variable Bayley Scales of Infant Development score: improvement by 18% at age 1 years.

Sample size: 60 patients: stratified into 3 groups to give power 0.85, alpha 0.05. Expect to accrue 2-4 patients per month.

ELIGIBILITY:
Inclusion Criteria:

* Neonates (<30 days) undergoing cardiac surgery with cardiopulmonary bypass will be enrolled.
* Inclusion criteria include patients with:

  * single ventricle: hypoplastic left heart syndrome or variant undergoing Norwood Stage I or Sano palliation (SV group);
  * patients with D-transposition of the great vessels with or without ventricular septal defect (VSD) undergoing arterial switch operation with VSD closure if needed (ASO group); and
  * patients with interrupted or hypoplastic aortic arch with intracardiac defects (VSD, ASD, or subaortic stenosis) who are undergoing complete 2- ventricle repair including aortic arch advancement(AAA group), any other 2 ventricle lesion scheduled for complex anatomic repair.

Exclusion Criteria:

* Gestational age less than 35 weeks at birth
* Weight less than 2 kg
* Known recognizable dysmorphic syndrome
* Surgery not requiring cardiopulmonary bypass
* Preoperative cardiac arrest requiring chest compressions for greater than 3 minutes
* Inability to enroll the patient greater than 12 hours preoperatively
* Aortic crossclamping is not used
* CPB times are anticipated to be less than 60 minutes
* A nadir temperature on bypass greater than 25° C is planned.
* Presence of known contraindications to EPO administration-sustained systolic blood pressure >100, hemoglobin .18 g/dL, known allergy to EPO or one of its components
* Platelet count >600,000 per dL, INR <0.8.
* Maternal history of major vascular thrombosis, or multiple fetal loss (3 or more spontaneous abortions).

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2006-09; Primary Completion 2012-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean B. Andropoulos, M.D., Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Kellert BA, McPherson RJ, Juul SE. A comparison of high-dose recombinant erythropoietin treatment regimens in brain-injured neonatal rats. Pediatr Res. 2007 Apr;61(4):451-5. doi: 10.1203/pdr.0b013e3180332cec. PMID 17515870
- [Background] McPherson RJ, Demers EJ, Juul SE. Safety of high-dose recombinant erythropoietin in a neonatal rat model. Neonatology. 2007;91(1):36-43. doi: 10.1159/000096969. Epub 2006 Nov 10. PMID 17344650
- [Background] Galli KK, Zimmerman RA, Jarvik GP, Wernovsky G, Kuypers MK, Clancy RR, Montenegro LM, Mahle WT, Newman MF, Saunders AM, Nicolson SC, Spray TL, Gaynor JW. Periventricular leukomalacia is common after neonatal cardiac surgery. J Thorac Cardiovasc Surg. 2004 Mar;127(3):692-704. doi: 10.1016/j.jtcvs.2003.09.053. PMID 15001897
- [Background] Andropoulos DB, Stayer SA, Diaz LK, Ramamoorthy C. Neurological monitoring for congenital heart surgery. Anesth Analg. 2004 Nov;99(5):1365-1375. doi: 10.1213/01.ANE.0000134808.52676.4D. PMID 15502032
- [Background] Andropoulos DB, Stayer SA, McKenzie ED, Fraser CD Jr. Regional low-flow perfusion provides comparable blood flow and oxygenation to both cerebral hemispheres during neonatal aortic arch reconstruction. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1712-7. doi: 10.1016/s0022-5223(03)01027-4. PMID 14688677
- [Background] Maiese K, Li F, Chong ZZ. New avenues of exploration for erythropoietin. JAMA. 2005 Jan 5;293(1):90-5. doi: 10.1001/jama.293.1.90. PMID 15632341
- [Background] McQuillen PS, Barkovich AJ, Hamrick SE, Perez M, Ward P, Glidden DV, Azakie A, Karl T, Miller SP. Temporal and anatomic risk profile of brain injury with neonatal repair of congenital heart defects. Stroke. 2007 Feb;38(2 Suppl):736-41. doi: 10.1161/01.STR.0000247941.41234.90. PMID 17261728
- [Background] Chang YS, Mu D, Wendland M, Sheldon RA, Vexler ZS, McQuillen PS, Ferriero DM. Erythropoietin improves functional and histological outcome in neonatal stroke. Pediatr Res. 2005 Jul;58(1):106-11. doi: 10.1203/01.PDR.0000163616.89767.69. Epub 2005 May 5. PMID 15879287
- [Background] Ballweg JA, Wernovsky G, Gaynor JW. Neurodevelopmental outcomes following congenital heart surgery. Pediatr Cardiol. 2007 Mar-Apr;28(2):126-33. doi: 10.1007/s00246-006-1450-9. Epub 2007 Jan 29. PMID 17265108
- [Background] Karl TR, Hall S, Ford G, Kelly EA, Brizard CP, Mee RB, Weintraub RG, Cochrane AD, Glidden D. Arterial switch with full-flow cardiopulmonary bypass and limited circulatory arrest: neurodevelopmental outcome. J Thorac Cardiovasc Surg. 2004 Jan;127(1):213-22. doi: 10.1016/j.jtcvs.2003.06.001. PMID 14752433
- [Background] Wypij D, Newburger JW, Rappaport LA, duPlessis AJ, Jonas RA, Wernovsky G, Lin M, Bellinger DC. The effect of duration of deep hypothermic circulatory arrest in infant heart surgery on late neurodevelopment: the Boston Circulatory Arrest Trial. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1397-403. doi: 10.1016/s0022-5223(03)00940-1. PMID 14666011
- [Background] Zhu C, Kang W, Xu F, Cheng X, Zhang Z, Jia L, Ji L, Guo X, Xiong H, Simbruner G, Blomgren K, Wang X. Erythropoietin improved neurologic outcomes in newborns with hypoxic-ischemic encephalopathy. Pediatrics. 2009 Aug;124(2):e218-26. doi: 10.1542/peds.2008-3553. Epub 2009 Jul 27. PMID 19651565
- [Background] Andropoulos DB, Mizrahi EM, Hrachovy RA, Stayer SA, Stark AR, Heinle JS, McKenzie ED, Dickerson HA, Meador MR, Fraser CD Jr. Electroencephalographic seizures after neonatal cardiac surgery with high-flow cardiopulmonary bypass. Anesth Analg. 2010 Jun 1;110(6):1680-5. doi: 10.1213/ANE.0b013e3181dd5a58. Epub 2010 Apr 30. PMID 20435942
- [Background] Andropoulos DB, Hunter JV, Nelson DP, Stayer SA, Stark AR, McKenzie ED, Heinle JS, Graves DE, Fraser CD Jr. Brain immaturity is associated with brain injury before and after neonatal cardiac surgery with high-flow bypass and cerebral oxygenation monitoring. J Thorac Cardiovasc Surg. 2010 Mar;139(3):543-56. doi: 10.1016/j.jtcvs.2009.08.022. Epub 2009 Nov 11. PMID 19909994
- [Background] McPherson RJ, Juul SE. Erythropoietin for infants with hypoxic-ischemic encephalopathy. Curr Opin Pediatr. 2010 Apr;22(2):139-45. doi: 10.1097/MOP.0b013e328336eb57. PMID 20090525
- [Background] Juul SE, McPherson RJ, Bauer LA, Ledbetter KJ, Gleason CA, Mayock DE. A phase I/II trial of high-dose erythropoietin in extremely low birth weight infants: pharmacokinetics and safety. Pediatrics. 2008 Aug;122(2):383-91. doi: 10.1542/peds.2007-2711. PMID 18676557
- [Background] Fauchere JC, Dame C, Vonthein R, Koller B, Arri S, Wolf M, Bucher HU. An approach to using recombinant erythropoietin for neuroprotection in very preterm infants. Pediatrics. 2008 Aug;122(2):375-82. doi: 10.1542/peds.2007-2591. PMID 18676556
- [Background] Brown MS, Eichorst D, Lala-Black B, Gonzalez R. Higher cumulative doses of erythropoietin and developmental outcomes in preterm infants. Pediatrics. 2009 Oct;124(4):e681-7. doi: 10.1542/peds.2008-2701. Epub 2009 Sep 28. PMID 19786428
- [Result] Andropoulos DB, Brady K, Easley RB, Dickerson HA, Voigt RG, Shekerdemian LS, Meador MR, Eisenman CA, Hunter JV, Turcich M, Rivera C, McKenzie ED, Heinle JS, Fraser CD Jr. Erythropoietin neuroprotection in neonatal cardiac surgery: a phase I/II safety and efficacy trial. J Thorac Cardiovasc Surg. 2013 Jul;146(1):124-31. doi: 10.1016/j.jtcvs.2012.09.046. Epub 2012 Oct 23. PMID 23102686
- See also: Texas Children's Hospital Web Site — http://TexasChildrensHospital.org
- See also: Baylor College of Medicine Web Site — http://www.bcm.edu
- See also: Congenital Cardiac Anesthesia Society Web Page — http://www.pedsanesthesia.org/ccas/
- See also: American Heart Association Web Page--Congenital Heart Disease — http://www.americanheart.org/children.
- See also: National Institutes of Health: National Institute of Child Health and Developement Web Site — http://www.nichd.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from September 2006 to February 2011 in the Texas Children's Hospital Heart Center NICU and CVICU.
Pre-assignment Details: 357 assessed for eligibility; 253 did not meet inclusion criteria. 42 subjects that eligible but consent not obtained (24 declined, 2 enrolled in another study, 16 investigator not available for consent or patient lived too far away). 62 consented, enrolled, received 1 dose EPO, but intended surgery not done on 3 subjects (no CPB); leaving 59.
Groups:
- Control Group.: Patients randomized to receive 3 doses of normal saline control.
  Normal saline: Normal saline placebo in 3 doses:dose 1. 12-72 hours preoperatively, dose 2. Postoperative day #1, 48 hours after separating from cardiopulmonary bypass, and dose 3. postoperative day #3, 48 hours after dose #2.
  .
Period: Overall Study
Arm/Group | EPO Group | Control Group.
Started | 35 (3 did not have intended surgery; 28 had all 3 doses; 4 had 1 dose but no more due to delayed surgery) | 27 (25 had 3 doses; 1 had 1 dose due to rash; 1 had 2 doses and 1 dose of EPO due to pharmacy error)
Clinical Data Collection &Pre/Postop MRI | 32 (3 not having intended surgery are subtracted from original 35 subjects, leaving 32) | 27
Completed | 22 (Competed 12 month neurodevelopmental exam, which are the only results published at this time.) | 20 (Competed 12 month neurodevelopmental exam, which are the only results published at this time.)
Not Completed | 13 | 7
Not completed — Did not have intended surgery | 3 | 0
Not completed — Death | 3 | 3
Not completed — Withdrawal by Subject | 7 | 4

BASELINE CHARACTERISTICS:
Population: These were the number of subjects followed for the intention-to-treat analysis because they received at least one dose of study drug/placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | EPO Group | Control Group. | Total
Number analyzed (Participants) | 32 | 27 | 59
Age, Continuous [Mean (Standard Deviation); unit: days] — Age at inclusion surgery
  days | 8.94 (5.35) | 8.12 (4.09) | 8.58 (4.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 16 | 16 | 32
Cardiac diagnosis [Number; unit: participants]
  Hypoplastic Left Heart Syndrome (HLHS) | 16 | 10 | 26
  (D-Transposition of the Great Arteries (D-TGA) | 9 | 12 | 21
  Aortic Arch & Ventricular Septal Defect/Other | 7 | 5 | 12
Any preoperative MRI injury [Number; unit: participants]
  Injury | 13 | 9 | 22
  No Injury | 19 | 18 | 37
New postoperative MRI injury [Number; unit: participants]
  Injury | 13 | 13 | 26
  No Injury | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Relative Difference in Total Maturity Score (TMS) From Preoperative Brain MRI to 7 Day Postoperative MRI
Description: TMS is a measure of developmental maturity of the brain as assessed from T1 and T2-weighted images, grading myelination, cortical infolding, involution of the germinal matrix, and presence of bands of migrating glial cells. The brain MRIs were reviewed for infarction, hemorrhage, white matter injury (WMI), or dural sinovenous thrombosis (DVST). Injuries in each category are scored 0 for none, 1 for mild, 2 for moderate, 3 for severe. The score in each category is then multiplied by a proposed outcome significance multiplier. A total injury score of 0 signifies no injury, 1-5 a mild injury, 6-10 a moderate injury, and >10 a severe injury. Range of scores is 0 - 51. Lower scores indicate less injury.
  The results present the relative difference of this score between the pre- and post-operative MRI. This was calculated as ((Post-operative MRI TMS - Pre-operative MRI TMS) / (Absolute(Pre-operative MRI TMS)) ). The proportion is then converted into a percentage.
Time Frame: 7 days postoperatively.
Population: Preoperative and postoperative MRIs were available to be scored on 33 subjects.
Measure: Mean (Full Range); unit: Percentage
Groups:
- Placebo Group: Patients randomized to receive 3 doses of normal saline control.
  Normal saline: Normal saline placebo in 3 doses:dose 1. 12-72 hours preoperatively, dose 2. Postoperative day #1, 48 hours after separating from cardiopulmonary bypass, and dose 3. postoperative day #3, 48 hours after dose #2.
  .
Arm/Group | EPO Group | Placebo Group
Number analyzed (Participants) | 17 | 16
Percentage | 12.1 [0 to 37.5] | 9.44 [0 to 30]

2. Primary Outcome: Scores on Bayley Scales of Infant Development III at Age 1 Years.
Description: 3 domains of the Bayley Scales of Infant Development III: Cognitive, Language and Motor Minimum score = 45, maximum score = 155; Population mean = 100, SD = 15; Higher scores are indicative of better outcomes Language scores are reflective of receptive communication and expressive communication subscales. Motor scores are reflective of fine motor and gross motor subscales.
Time Frame: 1 year postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EPO 1000 Units/kg QDx3: Original dose of 1000 units/kg every day for 3 doses
- EPO 500 Units/kg QODx3: Revised dose after FDA clinical hold removed of EPO 500 units/kg every other day for 3 doses
- Placebo: Normal saline control
Arm/Group | EPO 1000 Units/kg QDx3 | EPO 500 Units/kg QODx3 | Placebo
Number analyzed (Participants) | 11 | 11 | 20
units on a scale
  12-Month BSID-III Cognitive | 101.4 (16.9) | 100.9 (10.2) | 106.3 (10.7)
  12-Month BSID-III Language | 85.0 (16.3) | 92.0 (7.3) | 92.4 (12.4)
  12-Month BSID-III Motor | 89.3 (15.7) | 90.5 (8.6) | 92.6 (14.1)

3. Secondary Outcome: EEG Seizure Burden in the First 72 Postoperative Hours. (Total Minutes of EEG Seizures).
Time Frame: 72 hours postoperatively.
Measure: Mean (Full Range); unit: minutes
Arm/Group | EPO Group | Placebo Group
Number analyzed (Participants) | 32 | 27
minutes | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Pharmacokinetics of High Dose Erythropoetin: 7 Erythropoetin Levels in First 24 Hours After First Dose (Maximum EPO Plasma Concentration)
Time Frame: 24 hours after first EPO dose.
Population: Three patients had pharmacokinetic data obtained; 1 placebo and 2 patients who received EPO 1000 units/kg. Pharmacokinetic modeling was not performed because of these small patient numbers; however, maximum EPO plasma concentrations were measured in the EPO group. Outcome does not apply to the Placebo group and as such they were not analyzed.
Measure: Mean (Full Range); unit: mIU/mL
Arm/Group | EPO Group | Placebo Group
Number analyzed (Participants) | 2 | 0
mIU/mL | 6931 [5447 to 8415] |

ADVERSE EVENTS:
Arm/Group | EPO Group | Control Group.
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/27
Other Adverse Events (participants affected / at risk) | 4/35 | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPO Group (N=35) | Control Group. (N=27)
Postoperative dural sinovenous thrombosis (Nervous system disorders) | 3 (3) | 3 (3) — As evidenced by MRI exam
Clinical seizures (Nervous system disorders) | 1 (1) | 0 (0) — Clinical seizures diagnosed by physician exam
New cerebral infarction adjacent to thrombosis on postop MRI (Nervous system disorders) | 1 (1) | 0 (0) — New cerebral infarction adjuacent to thrombosis on postop MRI
Postop ECMO (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac arrest and subsequent ECMO

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes